CLINICAL TRIAL: NCT06429904
Title: A Prospective, Single Arm Study of Nimotuzumab Combined With NALIRIFOX in the Treatment of Locally Advanced Pancreatic Cancer
Brief Title: Nimotuzumab Plus NALIRIFOX in Locally Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-PC-29
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Nimotuzumab; locally advanced pancreatic cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab combined with NALIRIFOX (Experimental): Nimotuzumab combined with NALIRIFOX in the treatment of locally advanced pancreatic cancer
  Interventions: Drug: Nimotuzumab+ NALIRIFOX

INTERVENTIONS:
Drug: Nimotuzumab+ NALIRIFOX — Drug: Nimotuzumab Patients will receive Nimotuzumab 400 mg weekly or Nimotuzumab 600mg, 600mg, 400mg on Day 1, 8, 15, respectively, 28 days as a cycle, up to 6 cycles.
  Other Names: h-R3
  Drug: NALIRIFOX Patients will receive NALIRIFOX (liposomal irinotecan 50 mg/m2, oxaliplatin 60 mg/m2, leucovorin 400 mg/m2, and fluorouracil 2400 mg/m2, administered sequentially as a continuous intravenous infusion over 46 h) on days 1 and 15 of a 28-day cycle, up to 6 cycles.
  Other Names: NALIRIFOX

SUMMARY:
This is a prospective, open-label, single arm clinical study. The main purpose of the study is to evaluate the clinical efficacy and safety of Nimotuzumab combined with NALIRIFOX in the treatment of locally advanced pancreatic cancer (LAPC).

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, open-label, single arm study to evaluate the clinical efficacy and safety of Nimotuzumab combined with NALIRIFOX in the treatment of locally advanced pancreatic cancer (LAPC). Patients will receive Nimotuzumab plus NALIRIFOX as conversion therapy, and imaging assessments (according to RECIST V.1.1 criteria) will be performed every two cycles (every two months) of conversion therapy. The resectability of the primary pancreatic lesion will be judged based on NCCN guidelines and will be determined by a multidisciplinary team of experts. The main endpoint is overall survival (OS). Additional end points included resection rates, progression-free survival (PFS), objective response rate (ORR), safety, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender unlimited;
2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
3. Locally advanced pancreatic cancer, no evidence of distant metastasis as demonstrated by imaging;
4. Receive nimotuzumab and NALIRIFOX for voluntary, and patients can tolerate NALIRIFOX by researcher's evaluation;
5. No prior tumor systemic therapy.
6. Measurable disease according to RECIST criteria v1.1;
7. Adequate organ and bone marrow function, defined as follows: hemoglobin≥9.0 g/dL; absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥100×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
9. Postoperative survival was expected to be ≥3 months;
10. Fertile subjects are willing to take contraceptive measures during the study period.
11. Good compliance and signed informed consent voluntarily.

Exclusion Criteria:

1. Refuse chemotherapy or surgery;
2. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
3. Accompanied by other serious diseases, including but not limited to: compensatory heart failure (NYHA grade III and IV), unstable angina, poorly controlled arrhythmias, uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); active infections; unmanageable diabetes mellitus; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; gastric outlet obstruction; Respiratory insufficiency;
4. Undergone major surgery within 30 days;
5. Use of EGFR-mab or EGFR-TKI within 30 days;
6. Known allergy to prescription or any component of the prescription used in this study;
7. With HIV, HPV, or syphilis infection, or active hepatitis (hepatitis B, hepatitis C)
8. Other reasons that are not suitable to participate in this study according to the researcher's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | Up to 24 months
  The time from the beginning of treatment to death due to any cause.

SECONDARY OUTCOMES:
resection rate | Up to 24 months
  The proportion of patients who underwent surgery.
progression-free survival (PFS) | Up to 24 months
  PFS, defined as the time from the beginning of treatment to disease progression or all-cause death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Objective response rate (ORR) | Up to 12 months
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
tumor-related markers | Up to 24 months
  To explore the influence of tumor-related markers such as CA199 and EGFR on prognosis.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No